CLINICAL TRIAL: NCT01059461
Title: Phase 2 Nerve Growth Factor (Cerebrolysin®) for Treatment of Neonatal Hypoxic Ischemic Encephalopathy
Brief Title: Study of Cerebrolysin for Treatment of Infants With History of Neonatal Hypoxic Ischemic Encephalopathy
Acronym: CerebroHIE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahar M.A. Hassanein, MD (Other)
Responsible Party: Sponsor-Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Children's Hospital, Faculty of Medicine, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB 00006379
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Hypoxic Ischemic Encephalopathy (HIE); Perinatal Asphyxia; Nerve growth factor; Cerebrolysin; Cerebral palsy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Hereditary Sensory and Autonomic Neuropathies; Cerebral Palsy | interventions — cerebrolysin; Nerve Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cerebrolysin®, neuroregeneration (Experimental): Injection of cerebrolysin® 0.1ml/kg IM twice weekly for 10 injections after discharge from NICU (postneonatal)
  Interventions: Drug: Cerebrolysin®

INTERVENTIONS:
Drug: Cerebrolysin® — injection of cerebrolysin® 0.1ml/kg IM twice weekly for 10 injections after discharge from NICU (postneonatal)
  Other Names: Nerve Growth Factor

SUMMARY:
The purpose of this study is to determine whether nerve growth factor (cerebrolysin®) therapy will improve the psychomotor outcome in infants with moderate and severe hypoxic ischemic encephalopathy after hospital discharge.

DETAILED DESCRIPTION:
Infants with perinatal history of moderate to severe Hypoxic ischemic encephalopathy HIE will receive 10 injections of cerebrolysin IM. Assessment of neurodevelopment will be done before , 3 and 6 months after therapy

ELIGIBILITY:
*Inclusion Criteria: Infant aged 3-6 months with perinatal history of moderate or severe HIE collected from his NICU's file. Criteria of neonatal asphyxia and encephalopathy according to the American College of Obstetricians and Gynecologist and American Academy of Pediatrics, metabolic acidosis with a cord pH of 7.0 or less or a base deficit of at least 12 mmol/L, early onset of encephalopathy, and multisystem organ dysfunction with exclusion of other possible causes for findings.

Criteria of neonatal asphyxia:

* Full term neonate more than 36 weeks of gestation
* pH of 7.0 or less or a base deficit of 16 mmol per liter or more in a sample of umbilical-cord blood or any blood during the first hour after birth.
* If, during this interval, a pH is between 7.01 and 7.15, a base deficit is between 10 and 15.9 mmol per liter, or a blood gas is not available, additional criteria are required. These includes an acute perinatal event (e.g., late or variable decelerations, cord prolapse, cord rupture, uterine rupture, maternal trauma, hemorrhage, or cardiorespiratory arrest) and either a 10-minute Apgar score of 5 or less or assisted ventilation initiates at birth and continues for at least 10 minutes.

Criteria of neonatal encephalopathy according to Sarnat and Sarnat. Presence of one or more signs in at least three of the following six categories:

* level of consciousness.
* spontaneous activity.
* posture.
* tone.
* primitive reflexes (suck or Moro.
* autonomic nervous system (pupils, heart rate, or respiration). The number of moderate or severe signs determined the extent of encephalopathy; if signs were equally distributed, the designation was based on the level of consciousness.

  *Exclusion Criteria:
* Severe intrauterine growth retardation.
* Congenital malformations.
* Suspected inborn error of metabolism.
* Suspected inherited neurologic disease.
* Intracranial hemorrhage
* Meningitis

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Side effects during cerebrolysin therapy (one course). | 3 months
  weekly physical , neurological examination and parents' reported fever or convulsion during cerebrolysin injection course (10 injections).

SECONDARY OUTCOMES:
Neurodevelopmental follow up after 6 and 9 months of cerebrolysin injection. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MA Hassanein, MD, Principal Investigator — Children's Hospital, Faculty of Medicine, Ain Shams University
Locations (2):
- Egypt (2):
  - Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate
  - Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo